CLINICAL TRIAL: NCT00652704
Title: Randomized, Open-Label, 3-Way Crossover, Comparative Bioavailability Study of Par's and Oclassen's (Monodox) Doxycycline Monohydrate Capsules Administered as 1 x 100 mg Capsule in Healthy Adult Males Under Fasting and Fed Conditions
Brief Title: Bioavailability Study of Doxycycline Monohydrate Capsules and Monodox Under Fasting and Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Par Pharmaceutical, Inc. (Industry)
Collaborators: Anapharm (Industry)
Responsible Party: Alfred Elvin/Director of Biopharmaceutics, Par Pharmaceutical, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 99062
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: To Determine Bioequivalence Under Fed Conditions
Keywords: Bioequivalence; Doxycycline Monohydrate; Fed
MeSH Terms: conditions — Lecithin Cholesterol Acyltransferase Deficiency | interventions — Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): Subjects received the test product, Doxycycline Monohydrate Capsules (Par) under fed conditions
  Interventions: Drug: Doxycycline monohydrate
- B (Active Comparator): Subjects received the reference product, Monodox (Oclassen) under fed conditions
  Interventions: Drug: Monodox
- C (Experimental): Subjects received the test product, Doxycycline Monohydrate Capsules (Par) under fasting conditions
  Interventions: Drug: Doxycycline Monohydrate

INTERVENTIONS:
Drug: Doxycycline monohydrate — Capsules, 100 mg, fed
  Other Names: Monodox
  Arms: A
Drug: Monodox — Capsules, 100 mg, fed
  Other Names: Doxycycline Monohydrate
  Arms: B
Drug: Doxycycline Monohydrate — Capsules, 100 mg, fasting
  Other Names: Monodox
  Arms: C

SUMMARY:
To compare the rate and extent of absorption of doxycycline monohydrate capsules equivalent to 100 mg doxycycline (Par) versus Monodox (Oclassen Pharmaceuticals)

DETAILED DESCRIPTION:
To compare the rate and extent of absorption of doxycycline monohydrate capsules equivalent to 100 mg doxycycline by Par Pharmaceutical Inc., USA (test) versus Monodox by Oclassen Pharmaceuticals, Inc., USA (reference) administered as a 1 x 100 mg capsule under fasting and fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be males, non-smokers
* Between 18 and 55 years of age
* Subjects weight will be within 15% of their ideal body weight, based on Table of "Desirable Weight of Adults", Metropolitan Life Insurance Company, 1983
* Subjects should read, sign and date an Informed Consent Form prior to any study procedures
* Subjects must complete all screening procedures within 28 days prior to the administration of the study medication

Exclusion Criteria:

* Clinically significant anormalities found during medical screening
* Any clinically significant history of ongoing problems or problems known to interfere with the absorption, distribution, metabolism or excretion of drugs of drugs
* Clinically significant illnesses within 4 weeks of the administration of study medication
* Abnormal laboratory tests judged clinically significant
* ECG or vital sign abnormalities (clinically significant)
* History of allergic reactions to heparin
* Any food allergies, intolerances, restrictions, or special diet which in the opinion of the medical subinvestigator, contraindicates the subject's participation in the study
* History of severe allergies or hay fever
* Active asthma or bronchospasm
* Positive urine drug screen at screening
* Positive testing for hepatitis B, hepatitis C or HIV at screening
* Use of investigational drug or participation in an investigational study, within 30 days prior to administration of the study medication
* Recent donation of plasma (500 mL) within 7 days or recent donation or significant loss of whole blood (450 mL) within 56 days prior to the administration of the study medication
* History of significant alcohol abuse within six months of the screening visit or any indication of the regular use of more than two units of alcohol per day
* Recent history of drug abuse or use of illegal drugs: soft drugs (marijuana, pot) use within 3 months of the screening visit and hard drugs (cocaine, PCP, crack) use within 1 year of the screening visit
* Subjects who have taken prescription medication 14 days preceding administration of study medication or over-the-counter products 7 days preceding administration of study medication, except for topical products without systemic absorption
* Subjects who have taken any drugs known to induce or inhibit hepatic drug metabolism within 30 days prior to administration of the study medication
* Subjects who have undergone clinically significant surgery within 4 weeks prior to the administration of the study medication
* Any reason which, in the opinion of the medical subinvestigator, would prevent the subject from participating in the study

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 1999-07; Primary Completion 1999-09 (Actual); Study Completion 1999-09 (Actual)

PRIMARY OUTCOMES:
Rate and extent of absorption | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Eric Masson, Pharm.D., Principal Investigator — Anapharm
Locations (1):
- Anapharm, Inc., Sainte-Foy, Quebec, Canada